CLINICAL TRIAL: NCT03717077
Title: Effect of Learned Resourcefulness Intervention on Learned Resourcefulness, Caregiver Burden, Quality of Life for Older Family Caregivers
Brief Title: Learned Resourcefulness Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201801443B0C501
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Self-Control; Caregiver Burden; Quality of Life
MeSH Terms: conditions — Self-Control; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learned resourcefulness intervention (Experimental): The learned resourcefulness program includes: 1) Solving problem strategy, 2) Organizing daily actions, 3) Using self-regulation, 4) Reframing positive situations, 5) Changing negative self-thinking, 6) Exploring new thinking and skills. It is conducted one time per week.
  Interventions: Procedure: learned resourcefulness intervention
- Usual home care service (No Intervention): The control group maintains home care service

INTERVENTIONS:
Procedure: learned resourcefulness intervention — The LR program includes: 1) Solving problem strategy, 2) Organizing daily actions, 3) Using self-regulation, 4) Reframing positive situations, 5) Changing negative self-thinking, 6) Exploring new thinking and skills. It is conducted one time per week.
  Arms: Learned resourcefulness intervention

SUMMARY:
This study aimed to test the effects of a learned resourcefulness interveniton program on the learned resourcefulness, caregiver burden, quality of life for older family caregivers.

DETAILED DESCRIPTION:
A quasi-experimental trail will be used to test the effects of a learned resourcefulness intervention program on the learned resourcefulness, caregiver burden, quality of life for older family caregivers. Through the use of convenience sampling strategy, one teaching medical hospital with approximately 104 older family caregivers in southern Taiwan will be recruited and simple randomly assigned based on teaching medical hospital to a Learned resourcefulness intervention program experimental group or a wait-list control group. Participants in the experimental group will receive the learned resourcefulness intervention program led by researcher, one time per week, 50 minutes for one week, 10 minutes for these weeks; participants in the wait-list control group will continue to receive their home care service. One pre-test and two post-tests, all participants will assessed for learned resourcefulness, caregiver burden, quality of life at baseline, and at 5 and 9 weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 and above
* family caregivers of disabled adults who received home care service
* cognitively intact as assessed by SPMSQ score of 8 and above
* disabled adults will assessed by Barthel Index score of 60 and bellow
* able to answer questions

Exclusion Criteria:

* participants with severe mental disabilities

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Self-control as the learned resourcefulness measured by Rosenbaum's self control schedule | 9 weeks
  which is a 36-item scale, is used to measure the cognitive and problem-solving skills, the higher the score, the better a self-control of a person
Caregiver burden measured by caregiver burden scale | 9 weeks
  which is a 20-item scale by Lee and Wu, The total score ranges between 0 and 60, with a higher score representing a higher degree of burden.
Quality of life measured by EuroQol five dimension scale (ED-5Q) | 9 weeks
  The EuroQol five dimension scale (ED-5Q) developed by the EuroQol Group, the higher the score, the better the state of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Meng-Chun Chen (MCC), Chiayi City, Taiwan